CLINICAL TRIAL: NCT03151863
Title: Intranasal Dexmedetomidine for Procedural Pain Management in Elderly Adults in Palliative Care Setting: a Cross Over, Superiority, Double-blind, Controlled and Randomized Clinical Trial
Brief Title: Intranasal Dexmedetomidine for Procedural Pain Management in Elderly Adults in Palliative Care
Acronym: INDEX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of budget
Sponsor: Walid HABRE (Other)
Responsible Party: Sponsor-Investigator, Walid HABRE, Associate Professor, PhD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: INDEX_NDR
Record Dates: First submitted 2017-03-31; First posted 2017-05-12 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Analgesia; Sedation; Anxiolysis
Keywords: Dexmedetomidine; Opioids; Palliative Care; Elderly people; Nursing care; Analgesia; Sedation; Anxiolysis; Intranasal
MeSH Terms: conditions — Agnosia | interventions — Analgesics, Opioid; Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This two-sided, superiority, cross-over trial is based on a clinically relevant reduction (≥20%) of primary outcome (ECPA pain score >5) with the Dexmedetomidine treatment versus standard active control (opioids). It requires a sample size of 52 patients for a paired analysis with an intra-patient correlation of 50%.
  Type I error: 0.05 and type II error: 0.20. 25% of drop-out are expected. In consequence, 66 patients are required for the study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The nurse administers to the patient both subcutaneous and intranasal dose, however, one of the two is a placebo. The subcutaneous placebo and the subcutaneous opioids have the same packaging. Similar procedure is done for the intranasal compounds.
  Neither medical staff nor patient knows which analgesia is administered before this nursing care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioids, placebo (Active Comparator): One single dose of subcutaneous opioids and intranasal placebo (NaCl0.9%).
  Interventions: Drug: Opioids; Drug: Placebo
- Placebo, Dexmedetomidine (Experimental): One single dose of subcutaneous placebo (NaCl0.9%) and intranasal Dexmedetomidine 1.25ug/Kg
  Interventions: Drug: Dexmedetomidine; Drug: Placebo

INTERVENTIONS:
Drug: Opioids — The usual opioid treatment used for nursing care
  Other Names: Opioid prescribed to the patient on routine basis
  Arms: Opioids, placebo
Drug: Dexmedetomidine — Dexmedetomidine is provided intranasally
  Other Names: Dexdor
  Arms: Placebo, Dexmedetomidine
Drug: Placebo — Normal saline is either given subcutaneously or intranasally
  Other Names: Normal saline

SUMMARY:
Dexmedetomidine is allowed in Switzerland for intravenous (IV) medication in the intensive care unit in the adult patient. Its active molecule, Dexmedetomidine (Dex), is a selective and powerful α2-Adrenoreceptors (AR) agonist that shows the following complementary properties: anxiolytic, sedative and analgesic. Moreover, it displays interesting cardiovascular, respiratory and neuropsychic safety and tolerance profiles.

There is increasing number of promising studies for the use of intranasal (IN) Dex in pediatric sedation due to its non-invasive nature, its efficiency and its rare secondary effects. However, there is currently no information in the literature on the use of IN Dex in elderly multi-medicated patients in palliative care.

In this end-of-life population, pain is controlled with administration of opioids. Procedures, such as nursing cares, can generate pain and anxiety to the patient. Preventive analgesia, subcutaneous (SC) opioids, is administered before the care. However, most of the time, this additional dose fails to relieve the patient from his pain. In SPdol observational study, 42% daily hygiene and comfort nursing care remained painful despite the administration of a preventive analgesia.

IN Dex seems to be a good candidate for non-invasive analgesia and sedation in patients admitted in palliative care before the nursing procedure.

In this study, the investigators compare the efficiency of IN Dex to the regular extradose of SC opioids for analgesia before daily nursing care on elderly patients in the palliative care unit.

The study design is a cross over, two-sided, superiority, double-blind, placebo-controlled and randomized clinical trial.

DETAILED DESCRIPTION:
Although necessary for patient wellbeing, nursing care procedures potentially produce discomfort, that should be addressed before the procedures begin. In palliative care setting, daily procedures include mobilisation, hygiene care, wound dressing changes, etc. Non-invasive and simple nursing care procedures may cause anxiety and pain that can lead to a refusal of care or an increased distress. The data on procedural pain prevalence are almost only available in pediatrics and are scarce in palliative care and geriatric population. However, the SPdol french study, conducted on elderly people with palliative situations, showed that 85% of procedural pain was related to daily hygiene and comfort care. Results indicate also that in 42%, this type of care remained painful despite preventive pharmacologic measures as opioids administration. Intensity of procedural pain associated with daily and hygiene care is expected to be moderate to severe and not related to presence or absence of pain before initiation of the procedure but to bad prognostic.

In the context of chronic health problems, comfort management pharmacological interventions to achieve analgesia, slight or conscious sedation during nursing care procedures must ideally combine the following properties:

* Rapid recovery and excellent cardiovascular and respiratory security profile;
* Be administrable in the regular place of care of the patient;
* Minimal requirement for medical surveillance in terms of time, equipment and staff;
* Reproducible inset and outset of the analgesic and anxiolytic effect;
* Easy to titrate;
* Convenient, little or non-invasive and administration route as painless as possible.

Dexmedetomidine is allowed in Switzerland for intravenous (IV) medication in the intensive care unit in the adult patient. It is indicated to obtain a level of sedation no deeper than that allowing a response to a verbal stimulus. Its active molecule, Dexmedetomidine (Dex) is a selective and powerful agonist of α2-adrenoreceptors (AR). This drug has come to be of growing interest in anesthesia and sedation field these last years in literature. Its pharmacological actions on the central nervous system consist in sedative, anesthetic, anxiolytic, analgesic action with good cardiovascular, respiratory and neuropsychic tolerance profile. The main possible secondary effect with IV Dex is bradycardia, due to decreased circulating epinephrine and norepinephrine levels observed with this drug.

Intranasal (IN) administration is an easy-to-use and more efficient alternative than placebo or other sedatives (Midazolam, Ketamine, Chloral) for the sedation of sensitive or less collaborative populations as children and young adults.

IN Dex applications described in the literature include analgesia and sedation for the realization of radiologic investigation, surgical procedures leading to pain and anxiety, dental care, endoscopy and electrochemotherapy, in combination with local anesthesia. IN Dex doses from 1 to 2µg/Kg in young adults and up to 4µg/Kg in children,have been shown to be effective for analgesia and sedation, in these contexts.

From a pharmacological point of view, the superiority of the IN way compared to the oral one has been demonstrated in pediatrics. In healthy adults volunteers IN Dex bioavailability is 82% after a short time (2.6 min on average). The plasmatic peak of concentration is reached after 30 min on average (Tmax range 15-60min). The onset of sedation occurs at 45 min, with a peak effect observed at 90 min.

There is increasing number of promising studies for the use of IN Dex for pediatric sedation due to its non-invasive nature, its efficiency and its rare secondary effects. However, there is currently no information in the literature on the use of IN Dex neither in elderly patients nor in palliative situations.

In end-of-life population, pain is controlled with a subcutaneous administration of opioids as preventive analgesia before nursing cares, when necessary. Most of the time, this supplementary dose fails to relieve the patient from his pain. In SPdol observational study, 42% daily hygiene and comfort nursing care remained painful despite the administration of a preventive analgesia. Opioids limitations to prevent procedural pain are probably linked to anxiety and global discomfort induced by nursing care that opioids alone cannot alleviate. IN Dex seems to be a good candidate for procedural pain comfort pharmacological management giving its analgesic, anxiolytic and sedative properties in old people admitted with palliative situations.

In this study the investigators compare the efficiency of IN Dex to the regular additional dose of opioids for analgesia, sedation and anxiolysis for daily nursing care on end-of-life elderly patients.

The population of interest is widely heterogeneous according to its disease and medication. Moreover the pain feeling is specific to each person. Therefore a cross-over design was chosen so the patient is his own control. Each patient participates to 2 nursing care procedures where he receives both SC and IN administration. However, each time only one treatment is active while the other one is a placebo. Ex : SC placebo and IN Dex.

After a period of wash-out (24 to 48h), the patient receives , on the next nursing care procedure, the complementary treatment combination (ex: SC opioids and IN placebo).

To minimize bias, randomization is done by the pharmacy, on the treatment sequence and the study is double-blinded. In case of inefficient analgesia, the patient receives a rescue dose of Dormicum, 0.05mg/Kg.

During each procedure the patient is monitored with validated tools for pain, anxiety, sedation, heart rate and oxygen saturation.

The sedation state of the patient is assessed up to 45 minutes after treatment administration. At 45 minutes, the peak effect of the drugs (opioids as well as Dex) is reached and the nursing care can start and lasts for 15 to 30 minutes. The patient is followed-up during two hours after the end of the care. The total procedure lasts for 3h30 total.

ELIGIBILITY:
Inclusion criteria

* Informed consent signed and dated by the patient or a next of kin;
* ≥65 years old patients;
* Admitted in the palliative medicine unit;
* Undergoing, minimum once per day, a nursing care procedure lasting between 15 and 30 minutes causing discomfort (anxiety, pain or both) and therefore requiring the administration of an extra dose of Morphine, Hydromorphone before the nursing care;
* Taking, on a regularly basis, one of the following opioids: Morphine, Hydromorphone, Buprenorphine, Fentanyl.

Exclusion criteria

* Known hypersensitivity or allergy to Dexmedetomidine or Midazolam;
* Fentanyl extra dose medication before nursing cares;
* Weight > 80Kg;
* Psychomotor agitation;
* Known bronchial aspiration risks : ileus, vomiting, nausea, clinically relevant gastrooesophageal reflux;
* Known respiratory distress risk: recent need to be ventilated in Intensive Care Unit setting (<7 days), recent change or degradation of the respiratory status (<2 days) with apneas or tachypnea (>20/min), or known sleep apnea without non invasive ventilation; contraindication for nasal drug administration (ex. nasal tumour obstruction);
* Known cardiac risk : recent cardiac decompensation (<7 days) ; known life threatening or severe heart rate disorders ; bradycardia <60 bpm or known level II or III atrioventricular block without pacemaker ; hypotension with systolic blood pressure less or equal to 100 mmHg; Digoxine treatment;
* Known acute cerebrovascular disease or recent stroke (<1month);
* Already enrolled in another study or previous enrolment into the current study;
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Total score for ECPA over 5 | Minutes 35
  To assess the pain of the patient, a nurse will use the ECPA scale (Elderly Pain Caring Assessment). This is a validated tool to assess pain and anxiety intensity with 8 items based on the behaviour of the non-communicating elder person. The scale is divided in two: the first part is used for the pain assessment before the care while the second part assesses the pain during the care.
  The minimum score is 0. The maximum score is 32. One to five minutes are needed to do the evaluation depending on the experience of the observer.
  The pain is assessed 5 minutes before the care and then continuously during the care. When the total score between "before" and "during the care" exceeds 5, the patient is considered as having pain.

SECONDARY OUTCOMES:
Time to reach a level of sedation of mOAA less or equal to 4 before the care | Minutes 45
  The modified Observer's Assessment of Alertness/Sedation Scale (mOAA/S) is a validated tool with 7 levels, easy and rapid to use. One minute is sufficient to complete the assessment. The sedation state is evaluated every 15 minutes between the time when the drug is administered and the start of the care.
Time to come back to the initial sedation state | Hour 2
  The initial sedation state is evaluated with the mOAA/S scale before the administration of the drugs. After the end of the care, the sedation state of the patient is assessed every 30 minutes until he reaches his initial sedation state within maximum 2h.
anxiety | Minutes 35
  The anxiety (yes/no) is assessed with the ECPA scale. This scale includes anxiety items and will be used for this purpose also (see outcome 1).
Pain evolution | Minutes 90
  The pain is assessed by the patient himself using a Visual Analogue Scale

OTHER OUTCOMES:
Bradycardia | Hours 3 minutes 30
  Patient's heart rate is monitored during the whole procedure. Bradycardia (<60 beats per minutes) is one of the major risk observed with intravenous Dexmedetomidine.
Hypoxemia | Hours 3 minutes 30
  Patient's oxygen saturation is monitored during the whole procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Walid Habre, MD, PhD, Study Director — University of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
In case of request for a systematic review/meta-analysis, IPD can be shared after publication.

REFERENCES:
- [Derived] Dieudonne Rahm N, Zaccaria I, Gil Wey B, Pautex S, Habre W, Elia N. Intranasal Dexmedetomidine for Pain Management in Older Patients: A Cross-Over, Randomized, Double-Blinded, Active-Controlled Trial. Drugs Aging. 2023 Jun;40(6):527-538. doi: 10.1007/s40266-023-01027-3. Epub 2023 May 11. PMID 37170043